CLINICAL TRIAL: NCT00240019
Title: Maximizing the Benefit of RAS Blockade in Diabetic Nephropathy
Brief Title: Maximizing the Benefit of Renin-Angiotensin Blocking Drugs in Diabetic Renal Disease.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: R01-063011; R01DK063011 (NIH)
Record Dates: First submitted 2005-10-13; First posted 2005-10-17 (Estimated); Last update posted 2006-10-17 (Estimated); Status verified 2006-06

CONDITIONS: Diabetic Nephropathy
MeSH Terms: conditions — Diabetic Nephropathies

INTERVENTIONS:
Drug: Addition of furosemide 20 mg oral bid to baseline regimen

SUMMARY:
The angiotensin converting enzyme inhibitor drugs are now standard therapy for patients with diabetic nephropathy. The hypothesis of this study is that adding a diuretic agent (furosemide) will decrease the urine protein, which is a sign of disease, more than an angiotensin converting enzyme inhibitor alone.

ELIGIBILITY:
Inclusion Criteria:

proteinuria greater than 1 gram/day serum creatinine < 2.6 for men, < 2.0 for women

Exclusion Criteria:

blood pressure which cannot be controlled without a diuretic renal diseases other than diabetic nephropathy other disease which would alter renal function during 6 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2003-12; Study Completion 2006-04

PRIMARY OUTCOMES:
The amount of protein in the urine after 8 weeks of treatment.

SECONDARY OUTCOMES:
The estimated glomerular filtration rate after 8 weeks of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy W Meyer, MD, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - Kaiser Permanente of Northern California, Santa Clara and San Jose, Santa Clara, California
  - Stanford University Medical Center, Stanford, California